CLINICAL TRIAL: NCT05321368
Title: A Cardiometabolic Health Program Linked With Clinical-Community Support and Mobile Health Telemonitoring to Reduce Health Disparities
Acronym: LINKED-HEARTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00311760; P50MD017348 (NIH)
Record Dates: First submitted 2022-04-04; First posted 2022-04-11 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Hypertension; High Blood Pressure; Diabetes; Chronic Kidney Diseases
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LINKED-HEARTS Program (Experimental): Patients in the LINKED-HEARTS Program will be trained to measure their blood pressure with an Omron 10 series device using the Sphygmo telemonitoring app. The physician, pharmacist and Community Health Worker will have access to transmit data.
  Community Health Workers will provide education on managing blood pressure; reinforce positive blood pressure self-management behaviors; deliver knowledge and skills to promote healthy chronic conditions; assist with linking clinical and administrative services; and link participants with community resources.
  The study pharmacist will conduct telehealth visits, optimize pharmacologic therapy. The pharmacists will assess and address medication adherence to improve hypertension and diabetes control.
  Interventions: Behavioral: LINKED-HEARTS Program
- Enhanced Usual Care (No Intervention): Patients in the Enhanced Usual Care Arm, will receive care as usual from their primary care provider and will be trained to measure their blood pressure with an Omron 10 series device. The staff in each participating community health center practice will be trained in blood pressure measurement best practices.

INTERVENTIONS:
Behavioral: LINKED-HEARTS Program — The intervention arm will include training on home blood pressure monitoring, Sphygmo blood pressure telemonitoring app, Community Health Worker visit for education, counseling on lifestyles modification and Pharmacist to collaborate with other providers to optimize pharmacologic therapy to improve hypertension outcomes and with payors to ensure consistent access to drug therapy.
  Arms: LINKED-HEARTS Program

SUMMARY:
The LINKED- HEARTS Program is a multi-level project that intervenes at the practice level by linking home blood pressure monitoring (HBPM) with a telemonitoring platform (Sphygmo). The program incorporates team-based care by including community health workers (CHWs) and pharmacists to improve the outcomes of multiple chronic conditions (reduced blood pressure (BP), lower blood sugar, and improved kidney function). The LINKED-HEARTS Program will recruit a total of 600 adults with uncontrolled hypertension (BP ≥ 140/90 mm Hg) AND either type 2 diabetes or chronic kidney disease (CKD) across 16 community health centers or primary care practices serving high-risk adults. This cluster-randomized trial consists of two arms: (1) enhanced "usual care arm," wherein patients will be provided with Omron 10 series home BP monitors and will be managed by the patients' primary care clinicians as usual; and (2) the "intervention arm" which will integrate HBPM telemonitoring, a CHW intervention and provider-level interventions into the usual clinical care to improve BP control and provide support for self-management of chronic conditions. The study pharmacist will conduct telehealth, use the Sphygmo app and the Pharmacist Patient Care Process to collaborate with other providers to optimize pharmacologic therapy to improve hypertension outcomes and with payors to ensure consistent access to drug therapy.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age as of date of data extraction,
2. Self-identify as non-Hispanic white, non-Hispanic Black/African American and/or Hispanic,
3. Diagnosis of Hypertension (HTN) defined by International Classification of Diseases, Tenth code (ICD-10 code) and elevated systolic blood pressure (SBP) measure (≥140 mm Hg) on their most recent clinic visit.
4. Diagnosis of diabetes or chronic kidney disease (both defined by ICD-10 code), in addition to HTN
5. Receives primary medical care at one of the participating health systems
6. Have a Maryland and D.C. home address

Exclusion Criteria:

1. Age <18 years
2. Diagnosis of end-stage renal disease (ESRD) treated with dialysis
3. Serious medical condition which either limits life expectancy or requires active management (e.g., cancer)
4. Cognitive impairment or other condition preventing participation in the intervention
5. Planning to leave the practice or move out of the geographic area in 24 months
6. No longer consider the practice site their location for primary care
7. Unwillingness to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-10-21 (Estimated); Study Completion 2027-04-22 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure Control as assessed by percentage of participants with controlled Blood Pressure | 12 months
  Percent of patients with controlled Blood Pressure (<140/90 mm Hg).

SECONDARY OUTCOMES:
Change in Systolic Blood Pressure | Baseline and 12 months
  Change from baseline in mean systolic blood pressure in millimeters of mercury (mmHg).
Change in Diastolic blood pressure | Baseline and 12 months
  Change from baseline in diastolic blood pressure in mmHg.
Mean change in Hemoglobin A1c | Baseline and 12 months
  Mean change from baseline in hemoglobin A1c (percent) in patients with a diagnosis of diabetes.
Percent with Hemoglobin A1c < 7.0 | Baseline and 12 months
  Change from baseline in the percent with hemoglobin A1c < 7.0 in patients with a diagnosis of diabetes.
Change in Body Mass Index (BMI) | Baseline and 12 months
  Change from baseline in BMI (Kg/m^2).
Mean change in Estimated Glomerular Filtration Rate | Baseline and 12 months
  Mean change from baseline in Estimated Glomerular Filtration Rate.
Change in Health-Related Quality of Life as assessed by the PROMIS 29 | 12 months and 24 months
  This outcome will be measured using Patient-Reported Outcomes Measurement Information System®, (PROMIS) 29 Profile v. 2.0

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Commodore-Mensah, PhD, MSH, RN, Principal Investigator — JHU School Of Nursing
Locations (3):
- United States (3):
  - Unity Health Care, Washington D.C., District of Columbia
  - Johns Hopkins Community Physicians, Baltimore, Maryland
  - Choptank Community Health Systems, Denton, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Commodore-Mensah Y, Chen Y, Ogungbe O, Liu X, Metlock FE, Carson KA, Echouffo-Tcheugui JB, Ibe C, Crews D, Cooper LA, Himmelfarb CD. Design and rationale of the cardiometabolic health program linked with community health workers and mobile health telemonitoring to reduce health disparities (LINKED-HEARTS) program. Am Heart J. 2024 Sep;275:9-20. doi: 10.1016/j.ahj.2024.05.008. Epub 2024 May 15. PMID 38759910